CLINICAL TRIAL: NCT02116140
Title: Effects of Long Term Adaptive Servo Ventilation Therapy on Myocardial Energetics and Sympathetic Nerve Function in Heart Failure and Sleep Apnea. The AMEND Sub-study
Brief Title: ASV Effects on Myocardial Energetics and Sympathetic Nerve Function in Heart Failure and Sleep Apnea.
Acronym: AMEND
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ottawa Heart Institute Research Corporation (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 2011469-01; NA7158 (Other Grant/Funding Number: Heart & Stroke Foundation)
Record Dates: First submitted 2014-04-14; First posted 2014-04-16 (Estimated); Last update posted 2025-11-20 (Actual); Status verified 2025-11

CONDITIONS: Heart Failure; Obstructive Sleep Apnea; Central Sleep Apnea
Keywords: positron emission tomography; [11C]hydroxyephedrine (HED); [11C]acetate; Adaptive Servoventilation (ASV); Myocardial Energetics; work-metabolic index (WMI); Myocardial sympathetic neuron (SN) presynaptic function continuous positive airway pressure; heart rate variability; overnight polysomnogram; Plasma Norepinephrine; Urine Normetanephrine; Quality of Life
MeSH Terms: conditions — Heart Failure; Sleep Apnea, Obstructive; Sleep Apnea, Central | interventions — carbon-11 acetate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- [C11]Acetate HED PET (Experimental): AMEND is a single centre substudy of the ADVENT-HF trial. This substudy is a clinical physiologic proposal designed to determine the effects of long-term (6 months) ASV on cardiac energetics and SN function in patients with chronic stable HF and sleep apnea extending our previous evaluation of short-term CPAP in patients with OSA and HF.
  All subjects consenting to the ADVENT primary trial will be eligible to participate in the substudy.
  Substudy consenting patients will have [11C]acetate and [11C]HED PET imaging; HR variability; plasma norepinephrine (NE) levels, urine normetanephrine levels within 2 weeks of the sleep study. Baseline measurements will be repeated after 6 months in all patients.
  Interventions: Other: [C11]Acetate and HED PET

INTERVENTIONS:
Other: [C11]Acetate and HED PET

SUMMARY:
Obstructive sleep apnea (OSA), central sleep apnea (CSA) and heart failure (HF) are states of metabolic demand and sympathetic nervous system (SNS) activation. In patients with sleep apnea and HF, continuous positive airway pressure (CPAP) initially may reduce left ventricular (LV)stroke volume (SV) but subsequently improves and LV function. This may relate to an early beneficial effect on myocardial energetics through early reduction in metabolic demand that subsequently leads to improved efficiency of LV contraction. However, it is not clear whether long-term adaptive servo-ventilation (ASV) favorably affects cardiac energetics. Any such benefit may also relate to reduced sympathetic nervous system (SNS) activation. However its effect on myocardial SNS function is also not well studied.

In a pilot study we demonstrated early (6 week) beneficial effects of CPAP in patients with OSA and HF. The current proposal (AMEND) is a unique substudy of the recently funded ADVENT-HF trial (Adaptive Servo Ventilation for Therapy of Sleep Apnea in HeartFailure) (NCT01128816; CIHR; D. Bradley, PI).

We propose to evaluate the long-term (6 month) effects of ASV on daytime 1) oxidative metabolism; 2) the work metabolic index (WMI) as an estimate of mechanical efficiency; 3) myocardial sympathetic nerve (SN) pre-synaptic function; and 4) heart rate (HR) variability in patients with HF and coexisting OSA or CSA. In conjunction with echocardiographic measures of LV stroke work, positron emission tomography (PET) derived [11C] acetate kinetics will be used as a measure of oxidative metabolism, to determine the WMI. [11C] hydroxyephedrine (HED) retention will be used to measure cardiac SN pre-synaptic function.

Primary Hypotheses: In patients with chronic stable HF and CSA or OSA without excessive daytime sleepiness (EDS), long-term (6-month) ASV therapy yields:

1. Beneficial effects on daytime myocardial metabolism leading to a reduction in the rate of oxidative metabolism as measured by [11C]acetate kinetics using PET imaging;
2. Improvement in energy transduction from oxidative metabolism to stroke work as measured by an increase in the daytime work-metabolic index.

DETAILED DESCRIPTION:
DEFINITIONS Obstructive sleep apnea (OSA) is characterized by: episodes of partial or complete pharyngeal collapse leading to obstructive hypopnea and apnea during sleep. OSA often coexists with HF.

Central sleep apnea (CSA) is characterized by: reductions in central respiratory drive during sleep that leads to episodes of partial or complete cessation of airflow. CSA often co-exists with HF.

Continuous positive airway pressure(CPAP) delivers air through a nasal or oral interface to preserve upper airway patency. It is a treatment for symptomatic OSA or some patients with CSA.

Adaptive Servoventilation (ASV) is effective in alleviating OSA and CSA. It provides expiratory positive pressure to alleviate OSA, and inspiratory positive airway pressure to eliminate CSA.

Oxidative metabolism: utilization of substrates via the tricarboxylic acid cycle for Adenosine triphosphate (ATP) production; it is linked to myocardial oxygen consumption and can be measured with [11C]acetate PET.

The work-metabolic index (WMI) is the external work (minute-work) of the left ventricle corrected for the rate of oxidative metabolism and is an estimate of mechanical efficiency.

Myocardial sympathetic neuron (SN) presynaptic function is the measure of uptake and storage of neuronal catecholamines in the heart measured by [11C]hydroxyephedrine (HED) PET.

ELIGIBILITY:
This study (AMEND) is a single centre substudy of the ADVENT-HF trial (NCT01128816). ADVENT-HF is a RCT that will test the effects of ASV on morbidity and mortality in patients with HF and OSA or CSA.

The AMEND substudy is a clinical physiologic proposal designed to determine the effects of long-term (6 months) ASV on cardiac energetics and SN function in patients with chronic stable HF and sleep apnea extending our previous evaluation of short-term CPAP in patients with OSA and HF

Inclusion Criteria:

1. American Heart Association (AHA) Stages B, C and D heart failure due to ischemic, idiopathic or hypertensive causes with;
2. systolic dysfunction, ejection fraction (EF) ≤45% by echocardiography
3. optimal medical therapy conforming to the AHA guidelines (and for this proposal, stable therapy for >4 weeks)
4. sleep apnea with an Apnea/hypopnea Index ≥15, which will be divided into OSA (> 50% events obstructive), or CSA (> 50% of events central in nature)for patients with OSA, an Epworth Sleepiness Scale score of >10 and no or mild daytime sleepiness (by the International Classification of Sleep Disorders
5. age >18 years;
6. willingness to receive ASV therapy
7. informed consent

Exclusion Criteria:

1. Myocardial infarction, cardiac surgery or angioplasty within 3 months prior to enrollment,
2. listed for heart transplantation,
3. HF due to primary valvular heart disease,
4. pregnancy
5. current use of ASV or CPAP.
6. awaiting revascularization;
7. previous cardiac transplant;
8. life expectancy less than 6 months due to other co-morbidity;
9. a large transmural scar defined on previous perfusion imaging (severe resting perfusion defect (<50% uptake) occupying >25% of the LV);
10. concomitant treatment or use of: tricyclic antidepressants, cocaine or drugs which may alter catecholamine uptake.

For heart rate variability (HRV) analysis additional exclusions will include: a) a permanent pacemaker; b) atrial fibrillation; c) significant ventricular arrhythmia or sinus node dysfunction; patients may be excluded from HRV analysis and still be eligible for the sub-study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2012-07; Primary Completion 2026-06 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
ASV therapy yields a reduction in the rate of oxidative metabolism as measured by [11C]acetate kinetics using PET imaging in patients with HF, OSA and/or CSA | 6 months
ASV therapy yields an improvement in energy transduction from oxidative metabolism to stroke work as measured by an increase in the daytime work-metabolic index inpatients with HF, OSA and/or CSA. | 6 months

SECONDARY OUTCOMES:
ASV for CSA or OSA in patients with HF and sleep apnea will normalize daytime myocardial SN pre-synaptic function measured by [11C]HED retention on PET imaging, | 6 months
ASV for CSA or OSA in patients with HF and sleep apnea will normalize daytime sympathetic contributions to heart rate variability | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Rob S Beanlands, MD, Principal Investigator — Ottawa Heart Institute Research Corporation
Locations (1):
- University of Ottawa Heart Institute, Ottawa, Ontario, Canada

REFERENCES:
- [Background] Beanlands RS, Nahmias C, Gordon E, Coates G, deKemp R, Firnau G, Fallen E. The effects of beta(1)-blockade on oxidative metabolism and the metabolic cost of ventricular work in patients with left ventricular dysfunction: A double-blind, placebo-controlled, positron-emission tomography study. Circulation. 2000 Oct 24;102(17):2070-5. doi: 10.1161/01.cir.102.17.2070. PMID 11044422
- [Background] Yoshinaga K, Burwash IG, Leech JA, Haddad H, Johnson CB, deKemp RA, Garrard L, Chen L, Williams K, DaSilva JN, Beanlands RS. The effects of continuous positive airway pressure on myocardial energetics in patients with heart failure and obstructive sleep apnea. J Am Coll Cardiol. 2007 Jan 30;49(4):450-8. doi: 10.1016/j.jacc.2006.08.059. PMID 17258090